CLINICAL TRIAL: NCT05913544
Title: Short Integrative And Neurocognitive Therapy For Young Adults With Borderline Personality Disorder: a Study Model of Impulsivity Management
Brief Title: Short Integrative And Neurocognitive Therapy For Young Adults With Borderline Personality Disorder
Acronym: SINTYA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIMAO/2022-1/CE-01
Record Dates: First submitted 2023-05-22; First posted 2023-06-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-04

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SINTYA group (Experimental)
  Interventions: Other: SINTYA
- Control (No Intervention)

INTERVENTIONS:
Other: SINTYA — 10-week psychotherapy program consisting of a weekly 1h30 hour group therapy session plus 1 hour individual therapy session
  Arms: SINTYA group

SUMMARY:
Borderline personality disorder (BPD) is a severe, high-suicidal psychiatric disorder associated with impulsive, endangering behaviors. Young patients between 16 and 25 years old do not respond to traditional psychotherapies, which are often long and not adapted to their neurocognitive alterations linked to early trauma. The study authors hypothesize the SINTYA therapy program (one group session and one individual session weekly for 10 weeks) would reduce the level of impulsivity and clinical symptomatology (severity of the BPD; emotional regulation difficulties; dissociative symptoms; aggressiveness; ruminations; the number of self-destructive behaviors and suicidal acts; impulsive behaviors; level of suicide risk and hopelessness; the number of psychiatric hospitalizations and emergency visits for psychiatric reasons; and finally improving psychosocial functioning).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BPD according to DSM-5 criteria and BPQ-80 scale.
* High BPD severity level: ZAN-BPD (score ≥ 18/36).
* Understand, write and read French.
* Be able to understand the nature, purpose and methodology of the study and agree to cooperate during evaluations.
* Have signed the informed consent.
* For minor patients, have signed the parental consent by at least one holder of parental authority.

Exclusion Criteria:

* Refusal to participate.
* Existence of a neurological pathology or cerebral sequelae of organic origin which could affect neurocognitive performance.
* Intelligence quotient < 70.
* Lifetime diagnosis of schizoaffective disorder or schizophrenia (MINI-7).
* Previous or current participation in specific psychotherapy for BPD.
* Subject deprived of liberty (by judicial or administrative decision) and/or protected by law.
* Inclusion in another study including psychotherapy for the duration of the study.
* Inclusion in a drug RIPH1 study or in a REC study (European regulation of clinical trials) for the entire duration of the study.
* Subject in period of exclusion from another research protocol.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Variation in explicit impulsivity between groups | Baseline
  UPPS-S (Impulsive Behavior Scale Short version score)
Variation in explicit impulsivity between groups | Month 4
  UPPS-S (Impulsive Behavior Scale Short version score)

SECONDARY OUTCOMES:
Variation in explicit impulsivity between groups | Month 7
  UPPS-S (Impulsive Behavior Scale Short version score)
Variation in impulsiveness between groups | Baseline
  Barratt Impulsiveness Scale (BIS-11) (score out of 120)
Variation in impulsiveness between groups | Month 4
  Barratt Impulsiveness Scale (BIS-11) (score out of 120)
Variation in impulsiveness between groups | Month 7
  Barratt Impulsiveness Scale (BIS-11) (score out of 120)
BPD severity level between groups | Baseline
  Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) (score out of 36)
BPD severity level between groups | Month 4
  Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) (score out of 36)
BPD severity level between groups | Month 7
  Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) (score out of 36)
Emotional regulation capacities between groups | Baseline
  Difficulties in Emotion Regulation Scale (DERS-18)
Emotional regulation capacities between groups | Month 4
  Difficulties in Emotion Regulation Scale (DERS-18)
Emotional regulation capacities between groups | Month 7
  Difficulties in Emotion Regulation Scale (DERS-18)
Dissociative symptoms between groups | Baseline
  Dissociative Experiences Scale (DES): a score of 25 or higher is predictive of dissociative disorder
Dissociative symptoms between groups | Month 4
  Dissociative Experiences Scale (DES): a score of 25 or higher is predictive of dissociative disorder
Dissociative symptoms between groups | Month 7
  Dissociative Experiences Scale (DES): a score of 25 or higher is predictive of dissociative disorder
Aggression between groups | Baseline
  Aggression Questionnaire (AQ-12)
Aggression between groups | Month 4
  Aggression Questionnaire (AQ-12)
Aggression between groups | Month 7
  Aggression Questionnaire (AQ-12)
Ruminations between groups | Baseline
  Rumination Reflection Questionnaire (RRQ)
Ruminations between groups | Month 4
  Rumination Reflection Questionnaire (RRQ)
Ruminations between groups | Month 7
  Rumination Reflection Questionnaire (RRQ)
Number of self-destructive behaviors between groups | Baseline
  Number of self-destructive/self-mutilatory/parasuicidal acts reported by the patient in a clinical interview
Number of self-destructive behaviors between groups | Month 4
  Number of self-destructive/self-mutilatory/parasuicidal acts reported by the patient in a clinical interview
Number of self-destructive behaviors between groups | Month 7
  Number of self-destructive/self-mutilatory/parasuicidal acts reported by the patient in a clinical interview
Number of impulsive behaviors between groups | Baseline
  Number of impulsive behaviors (food, motor vehicles, sexual, drug-related)
Number of impulsive behaviors between groups | Month 4
  Number of impulsive behaviors (food, motor vehicles, sexual, drug-related)
Number of impulsive behaviors between groups | Month 7
  Number of impulsive behaviors (food, motor vehicles, sexual, drug-related)
Level of suicide risk between groups | Baseline
  Columbia-Suicide Severity Rating Scale (C-SSRS)
Level of suicide risk between groups | Month 4
  Columbia-Suicide Severity Rating Scale (C-SSRS)
Level of suicide risk between groups | Month 7
  Columbia-Suicide Severity Rating Scale (C-SSRS)
Number of psychiatric hospitalizations and emergency visits for psychiatric reasons between groups | 12 Months prior to inclusion
  Information taken from patient medical file
Number of psychiatric hospitalizations and emergency visits for psychiatric reasons between groups | Baseline
  Information taken from patient medical file
Number of psychiatric hospitalizations and emergency visits for psychiatric reasons between groups | Month 4
  Information taken from patient medical file
Number of psychiatric hospitalizations and emergency visits for psychiatric reasons between groups | Month 7
  Information taken from patient medical file
Psychosocial functioning between groups | Baseline
  Functional Assessment Staging Tool (FAST)
Psychosocial functioning between groups | Month 4
  Functional Assessment Staging Tool (FAST)
Psychosocial functioning between groups | Month 7
  Functional Assessment Staging Tool (FAST)
Implicit impulsivity between groups | Baseline
  Continuous Performance Test (CPT)
Implicit impulsivity between groups | Month 4
  Continuous Performance Test (CPT)
Implicit impulsivity between groups | Month 7
  Continuous Performance Test (CPT)
Neurocognitive evaluation of implicit impulsivity between groups | Baseline
  Emotional Stroop (SE) customized to the study
Neurocognitive evaluation of implicit impulsivity between groups | Month 4
  Emotional Stroop (SE) customized to the study
Neurocognitive evaluation of implicit impulsivity between groups | Month 7
  Emotional Stroop (SE) customized to the study
Risk taking between groups | Baseline
  Balloon Analogue Risk Task (BART)
Risk taking between groups | Month 4
  Balloon Analogue Risk Task (BART)
Risk taking between groups | Month 7
  Balloon Analogue Risk Task (BART)
Decision making under risk conditions between groups | Baseline
  Game Dice Task (GDT)
Decision making under risk conditions between groups | Month 4
  Game Dice Task (GDT)
Decision making under risk conditions between groups | Month 7
  Game Dice Task (GDT)

CONTACTS AND LOCATIONS:
Overall Officials: Clémentine Estric, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon publication
Access Criteria: The IPD will be made available to other researchers upon reasonable request to the corresponding author